CLINICAL TRIAL: NCT02036775
Title: An Open-label, Randomised, Multiple-dose, Three-period Crossover Study in Healthy Male and Female Volunteers to Characterise Pharmacokinetics and Assess the Relative Bioavailability of Two New Oral Formulations of Ambroxol Hydrochloride as Lasolvan® Prolonged-release Hard Capsules 75 mg and Lasolvan® Effervescent Tablets 60 mg Compared to Lasolvan® Tablets 30 mg.
Brief Title: Pharmacokinetics and Bioavailability Study of Lasolvan Hard Capsules and Effervescent Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18.510
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Results first posted 2015-05-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
MeSH Terms: interventions — Ambroxol

ARMS (6):
- Treatment sequence 1 (Experimental): Treatment 1, Washout 6 days, Reference product, Washout 6 days, Treatment 2
  Interventions: Drug: Lasolvan tablet; Drug: Lasolvan prolonged-released capsules; Drug: Lasolvan effervescent tablet
- Treatment sequence 2 (Experimental): Treatment 2, Washout period 6 days, Treatment 1, Washout 6 days, Reference product
  Interventions: Drug: Lasolvan tablet; Drug: Lasolvan effervescent tablet; Drug: Lasolvan prolonged-release hard capsule
- Treatment sequence 3 (Experimental): Reference product, Washout 6 days, Treatment 2, Washout 6 days, Treatment 1
  Interventions: Drug: Lasolvan effervescent tablet; Drug: Lasolvan tablet; Drug: Lasolvan prolonged-release hard capsule
- Treatment Sequence 4 (Experimental): Treatment 2, Washout 6 days, Reference product, Washout 6 days, Treatment 1
  Interventions: Drug: Lasolvan tablet; Drug: Lasolvan effervescent tablet; Drug: Lasolvan prolonged-release hard capsule
- Treatment sequence 5 (Experimental): Reference product, Washout 6 days, Treatment 1, Washout 6 days, Treatment 2
  Interventions: Drug: Lasolvan tablet; Drug: Lasolvan prolonged-release hard capsule; Drug: Lasolvan effervescent tablet
- Treatment Sequence 6 (Experimental): Treatment 1, Washout 6 days, Treatment 2, Washout 6 days, Reference product
  Interventions: Drug: Lasolvan tablet; Drug: Lasolvan effervescent tablet; Drug: Lasolvan prolonged-release hard capsule

INTERVENTIONS:
Drug: Lasolvan tablet — One Lasolvan tablet 30 mg twice daily for 5 days.
  Arms: Treatment sequence 1
Drug: Lasolvan tablet — One Lasolvan tablet 30 mg twice daily for 5 days.
  Arms: Treatment sequence 2
Drug: Lasolvan tablet — One Lasolvan tablet 30 mg twice daily for 5 days.
  Arms: Treatment Sequence 4
Drug: Lasolvan tablet — One Lasolvan tablet 30 mg twice daily for 5 days.
  Arms: Treatment Sequence 6
Drug: Lasolvan effervescent tablet — One-half Lasolvan effervescent tablet 60mg twice daily for 5 days.
  Arms: Treatment sequence 3
Drug: Lasolvan effervescent tablet — One-half Lasolvan effervescent tablet 60mg twice daily for 5 days.
  Arms: Treatment Sequence 4
Drug: Lasolvan effervescent tablet — One-half Lasolvan effervescent tablet 60mg twice daily for 5 days.
  Arms: Treatment Sequence 6
Drug: Lasolvan prolonged-release hard capsule — One Lasolvan prolonged-release hard capsule 75 mg once daily for 5 days
  Arms: Treatment Sequence 4
Drug: Lasolvan prolonged-release hard capsule — One Lasolvan prolonged-release hard capsule 75 mg once daily for 5 days
  Arms: Treatment Sequence 6
Drug: Lasolvan prolonged-released capsules — One Lasolvan prolonged-release hard capsule 75 mg once daily for 5 days
  Arms: Treatment sequence 1
Drug: Lasolvan tablet — One Lasolvan tablet 30 mg twice daily for 5 days.
  Arms: Treatment sequence 3
Drug: Lasolvan tablet — One Lasolvan tablet 30 mg twice daily for 5 days.
  Arms: Treatment sequence 5
Drug: Lasolvan prolonged-release hard capsule — One Lasolvan prolonged-release hard capsule 75 mg once daily for 5 days
  Arms: Treatment sequence 3
Drug: Lasolvan effervescent tablet — One-half Lasolvan effervescent tablet 60mg twice daily for 5 days.
  Arms: Treatment sequence 2
Drug: Lasolvan prolonged-release hard capsule — One Lasolvan prolonged-release hard capsule 75 mg once daily for 5 days
  Arms: Treatment sequence 5
Drug: Lasolvan prolonged-release hard capsule — One Lasolvan prolonged-release hard capsule 75 mg once daily for 5 days
  Arms: Treatment sequence 2
Drug: Lasolvan effervescent tablet — One-half Lasolvan effervescent tablet 60mg twice daily for 5 days.
  Arms: Treatment sequence 5
Drug: Lasolvan effervescent tablet — One-half Lasolvan effervescent tablet 60mg twice daily for 5 days.
  Arms: Treatment sequence 1

SUMMARY:
To characterise pharmacokinetics and assess the relative bioavailability of two new oral formulations of ambroxol hydrochloride as Lasolvan® prolonged-release hard capsules 75 mg and Lasolvan® effervescent tablets 60 mg compared to Lasolvan® tablets 30 mg

ELIGIBILITY:
Inclusion criteria:

* Given written informed consent for participation in the study.
* Male and female subjects aged 18-45, inclusive.
* Body mass index by Quetelet 18.50 - 24.99 kg/m2, inclusive.
* Judged by the investigator to be in good health as documented by the medical history, physical examination (including but may not be limited to an evaluation of the cardiovascular, gastrointestinal, and renal systems), vital signs assessments, 12-lead electrocardiogram (ECG), clinical laboratory assessments, and by general observations. Any abnormalities outside normal ranges for any clinical testing (laboratory tests, ECG, vital signs) can be repeated at the discretion of the investigator and judged to be not clinically significant for the study participation.
* Female subjects of childbearing potential who agree on using double-barrier contraception during the study. If female is postmenopausal (no menses for at least 1 year) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) she will be exempt from the requirement. In case of using oral contraceptives, they should be withdrawn at least 2 months before the study.
* Male subjects who agree on using effective contraception during the study (barrier contraceptive methods).

Exclusion criteria:

* Known hypersensitivity to ambroxol hydrochloride, or other constituents of the test and reference products.
* Known rare hereditary conditions (Stevens-Johnson syndrome, toxic epidermal necrolysis, galactose intolerance, Lapp-lactase deficiency, glucose-galactose malabsorption).
* Pregnancy or breastfeeding.
* Chronic hepatic, renal, cardiovascular, respiratory, gastrointestinal, neuroendocrine diseases and blood disorders.
* Positive results of blood tests for current infections (HIV, syphilis, hepatitis B or C).
* Surgery of gastro-intestinal tract (except of appendectomy) within the past 8 weeks.
* Acute infections occurred within 4 weeks before inclusion into the study.
* Regular drug intake within 2 weeks before inclusion into the study.
* Intake of systemic drugs known to affect cytochrome P450 system (induce or inhibit) within 4 weeks before inclusion into the study.
* Blood donation (greater or equal 450 ml) within 2 months before inclusion into the study.
* Alcohol intake greater than or equal to 10 units of alcohol per week (1 unit of alcohol equals one 50 ml single measure of whisky (ABV - alcohol by volume 40%), or 0.5 litre of beer (ABV 5%), or 200 ml glass of red wine (ABV 12%) or history of alcohol abuse, narcomania, or other drug abuse.
* A positive urine drug test (cannabis, benzodiazepines, barbiturates, opiates, cocaine, amphetamines) at screening and before the first dosing in each study period.
* A positive alcohol test at screening and before the first dosing in each study period
* Participation in another phase I clinical study within 3 months before inclusion into the study.
* Known lactose intolerance.
* Known phenylketonuria

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 18.510.2 Boehringer Ingelheim Investigational Site, Saint Petersburg, Russia

REFERENCES:
- [Derived] Ollier C, Sent U, Mesquita M, Michel MC. Pharmacokinetics of Ambroxol Sustained Release (Mucosolvan(R) Retard) Compared with Other Formulations in Healthy Volunteers. Pulm Ther. 2020 Jun;6(1):119-130. doi: 10.1007/s41030-020-00116-7. Epub 2020 May 5. PMID 32372294

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A randomised, open-label, three period, crossover study. Each subject received one treatment per treatment period. Each of the three treatment phases was 6 days long, where study drug was administered on day 1-5 during each treatment.
Groups:
- Lasolvan 75mg / Lasolvan 30mg / Lasolvan 60mg: Patients were administered three treatments in the following order:
  * One Lasolvan prolonged release hard capsule, 75mg, swallowed and taken with 200ml of boiled water once daily for 5 days
  * One Lasolvan tablet, 30mg, was taken with 200mL of boiled water twice daily for 5 days (reference treatment)
  * One-half Lasolvan effervescent tablet, 60mg, dissolved in 200mL of boiled water, taken twice daily for 5 days
- Lasolvan 60mg / Lasolvan 75mg / Lasolvan 30mg: Patients were administered three treatments in the following order:
  * One-half Lasolvan effervescent tablet, 60mg, dissolved in 200mL of boiled water, taken twice daily for 5 days
  * One Lasolvan prolonged release hard capsule, 75mg, swallowed and taken with 200ml of boiled water once daily for 5 days
  * One Lasolvan tablet, 30mg, was taken with 200mL of boiled water twice daily for 5 days (reference treatment)
- Lasolvan 30mg / Lasolvan 60mg / Lasolvan 75mg: Patients were administered three treatments in the following order:
  * One Lasolvan tablet, 30mg, was taken with 200mL of boiled water twice daily for 5 days (reference treatment)
  * One-half Lasolvan effervescent tablet, 60mg, dissolved in 200mL of boiled water, taken twice daily for 5 days
  * One Lasolvan prolonged release hard capsule, 75mg, swallowed and taken with 200ml of boiled water once daily for 5 days
- Lasolvan 60mg / Lasolvan 30mg / Lasolvan 75mg: Patients were administered three treatments in the following order:
  * One-half Lasolvan effervescent tablet, 60mg, dissolved in 200mL of boiled water, taken twice daily for 5 days
  * One Lasolvan tablet, 30mg, was taken with 200mL of boiled water twice daily for 5 days (reference treatment)
  * One Lasolvan prolonged release hard capsule, 75mg, swallowed and taken with 200ml of boiled water once daily for 5 days
- Lasolvan 30mg / Lasolvan 75mg / Lasolvan 60mg: Patients were administered three treatments in the following order:
  * One Lasolvan tablet, 30mg, was taken with 200mL of boiled water twice daily for 5 days (reference treatment)
  * One Lasolvan prolonged release hard capsule, 75mg, swallowed and taken with 200ml of boiled water once daily for 5 days
  * One-half Lasolvan effervescent tablet, 60mg, dissolved in 200mL of boiled water, taken twice daily for 5 days
- Lasolvan 75mg / Lasolvan 60mg / Lasolvan 30mg: Patients were administered three treatments in the following order:
  * One Lasolvan prolonged release hard capsule, 75mg, swallowed and taken with 200ml of boiled water once daily for 5 days
  * One-half Lasolvan effervescent tablet, 60mg, dissolved in 200mL of boiled water, taken twice daily for 5 days
  * One Lasolvan tablet, 30mg, was taken with 200mL of boiled water twice daily for 5 days (reference treatment)
Period: Treatment Period 1 (6 Days)
Arm/Group | Lasolvan 75mg / Lasolvan 30mg / Lasolvan 60mg | Lasolvan 60mg / Lasolvan 75mg / Lasolvan 30mg | Lasolvan 30mg / Lasolvan 60mg / Lasolvan 75mg | Lasolvan 60mg / Lasolvan 30mg / Lasolvan 75mg | Lasolvan 30mg / Lasolvan 75mg / Lasolvan 60mg | Lasolvan 75mg / Lasolvan 60mg / Lasolvan 30mg
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (6 Days)
Arm/Group | Lasolvan 75mg / Lasolvan 30mg / Lasolvan 60mg | Lasolvan 60mg / Lasolvan 75mg / Lasolvan 30mg | Lasolvan 30mg / Lasolvan 60mg / Lasolvan 75mg | Lasolvan 60mg / Lasolvan 30mg / Lasolvan 75mg | Lasolvan 30mg / Lasolvan 75mg / Lasolvan 60mg | Lasolvan 75mg / Lasolvan 60mg / Lasolvan 30mg
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment Period 3 (6 Days)
Arm/Group | Lasolvan 75mg / Lasolvan 30mg / Lasolvan 60mg | Lasolvan 60mg / Lasolvan 75mg / Lasolvan 30mg | Lasolvan 30mg / Lasolvan 60mg / Lasolvan 75mg | Lasolvan 60mg / Lasolvan 30mg / Lasolvan 75mg | Lasolvan 30mg / Lasolvan 75mg / Lasolvan 60mg | Lasolvan 75mg / Lasolvan 60mg / Lasolvan 30mg
Started | 4 | 4 | 4 | 4 | 4 | 3
Completed | 4 | 4 | 4 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set which included all subjects who had been dispensed study medication and were documented to have taken at least one dose of study medication.
Groups:
- Study Overall: A randomised, open-label, three period, crossover study. The three treatments administered were:
  * One Lasolvan prolonged release hard capsule, 75mg, swallowed and taken with 200ml of boiled water once daily for 5 days
  * One-half Lasolvan effervescent tablet, 60mg, dissolved in 200mL of boiled water, taken twice daily for 5 days
  * One Lasolvan tablet, 30mg, was taken with 200mL of boiled water twice daily for 5 days (reference treatment)
  Each subject received one treatment per treatment period. Each of the three treatment phases was 6 days long, where study drug was administered on day 1-5 during each treatment.
Arm/Group | Study Overall
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.04 (6.423)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to 24 h at Steady State
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 24 h at steady state (AUCss 0-24)
Time Frame: Pre-dose, 30min, 1h, 1h 30min, 2h, 3h, 4h, 5h, 6h, 7h 30min, 9h, 10h 30min, 12h, 14h, 17h, 20h, 24h after the morning dose for all treatments; also 15min, 45min, 12h 15min, 12h 30min, 12h 45min, 13h, 13h 30min, 15h, 16h for Lasolvan 60mg and Lasolvan 30mg
Population: Pharmacokinetic (PK) set relative bioavailability set (PK-BA set) which includes all subjects in the treated set who completed 3 periods and for whom the PK profiles in 3 periods could be adequately characterized in respect to at least 1 of the PK parameters of primary interest without important protocol violations relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Lasolvan 75mg: One Lasolvan prolonged release hard capsule, 75mg, swallowed and taken with 200ml of boiled water once daily for 5 days
- Lasolvan 60mg: One-half Lasolvan effervescent tablet, 60mg, dissolved in 200mL of boiled water, taken twice daily for 5 days
- Lasolvan 30mg: One Lasolvan tablet, 30mg, was taken with 200mL of boiled water twice daily for 5 days (reference treatment)
Arm/Group | Lasolvan 75mg | Lasolvan 60mg | Lasolvan 30mg
Number analyzed (Participants) | 23 | 23 | 23
ng*h/mL | 1182.084 (28.859) | 1110.095 (28.292) | 1070.909 (32.259)
Statistical Analysis 1: Comparison: Lasolvan 75mg vs Lasolvan 30mg; Test type: Non-Inferiority or Equivalence — The assessment of relative bioavailability without molar mass adjustment (dose adjustment) was based upon two-sided 90% confidence intervals (CIs) for the ratios of the geometric means (test divided by reference) of the area under the curve (AUCss 0-24) using an acceptance range of 80%-125%; Adjusted Geometric Mean Ratio (%) = 110.68, 90% CI 2-sided [99.84 to 122.69], Standard Deviation 20.42 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV(%))
Statistical Analysis 2: Comparison: Lasolvan 60mg vs Lasolvan 30mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Adjusted Geometric Mean Ratio (%) = 103.39, 90% CI 2-sided [96.54 to 110.74], Standard Deviation 13.52 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV(%))
Statistical Analysis 3: Comparison: Lasolvan 75mg vs Lasolvan 60mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Adjusted Geometric Mean Ratio (%) = 106.93, 90% CI 2-sided [100.29 to 114.02], Standard Deviation 12.65 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV(%))

2. Primary Outcome: Maximum Measured Concentration of the Analyte in Plasma at Steady State
Description: Maximum measured concentration of the analyte in plasma at steady state (Cmax ss)
Time Frame: as for outcome 1
Population: PK-BA set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lasolvan 75mg | Lasolvan 60mg | Lasolvan 30mg
Number analyzed (Participants) | 23 | 23 | 23
ng/mL | 73.510 (26.927) | 90.755 (34.426) | 87.289 (34.426)
Statistical Analysis 1: Comparison: Lasolvan 75mg vs Lasolvan 30mg; Test type: Non-Inferiority or Equivalence — The assessment of relative bioavailability without molar mass adjustment (dose adjustment) was based upon two-sided 90% confidence intervals (CIs) for the ratios of the geometric means (test divided by reference) of the peak concentration (Cmax ss) using an acceptance range of 75%-133%; Adjusted Geometric Mean Ratio (%) = 84.72, 90% CI 2-sided [76.96 to 93.25], Standard Deviation 19.01 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV(%))
Statistical Analysis 2: Comparison: Lasolvan 60mg vs Lasolvan 30mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Adjusted Geometric Mean Ratio (%) = 103.87, 90% CI 2-sided [95.22 to 113.31], Standard Deviation 17.19 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV(%))
Statistical Analysis 3: Comparison: Lasolvan 75mg vs Lasolvan 60mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Adjusted Geometric Mean Ratio (%) = 80.94, 90% CI 2-sided [73.92 to 88.62], Standard Deviation 17.95 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV(%))

3. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma at Steady State During 0-24 h, Adjusted to a Daily Dose of 60 mg
Description: Area under the concentration-time curve of the analyte in plasma at steady state during 0-24 h, adjusted to a daily dose of 60 mg (AUCss 0-24 norm)
Time Frame: as for outcome 1
Population: PK-BA set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Lasolvan 75mg | Lasolvan 60mg | Lasolvan 30mg
Number analyzed (Participants) | 23 | 23 | 23
ng*h/mL | 945.667 (28.859) | 1110.095 (28.292) | 1070.909 (32.259)
Statistical Analysis 1: Comparison: Lasolvan 75mg vs Lasolvan 30mg; Test type: Non-Inferiority or Equivalence — The assessment of relative bioavailability without molar mass adjustment (dose adjustment) was based upon two-sided 90% confidence intervals (CIs) for the ratios of the geometric means (test divided by reference) for the dose-adjusted total exposure (AUCss 0-24 norm) using an acceptance range of 80%-125%; Adjusted Geometric Mean Ratio (%) = 88.54, 90% CI 2-sided [79.87 to 98.15], Standard Deviation 20.42 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV(%))
Statistical Analysis 2: Comparison: Lasolvan 60mg vs Lasolvan 30mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Adjusted Geometric Mean Ratio (%) = 103.39, 90% CI 2-sided [96.54 to 110.74], Standard Deviation 13.52 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV(%))
Statistical Analysis 3: Comparison: Lasolvan 75mg vs Lasolvan 60mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Adjusted Geometric Mean Ratio (%) = 85.55, 90% CI 2-sided [80.23 to 91.22], Standard Deviation 12.65 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV(%))

4. Secondary Outcome: Rate of Absorption at Steady State (Cmax ss/AUCss 0-24)
Description: Metric which characterises the rate of absorption at steady state (Cmax ss/AUCss 0-24)
Time Frame: as for outcome 1
Population: PK-BA set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Lasolvan 75mg | Lasolvan 60mg | Lasolvan 30mg
Number analyzed (Participants) | 23 | 23 | 23
1/h | 0.062 (13.477) | 0.082 (14.568) | 0.082 (13.477)
Statistical Analysis 1: Comparison: Lasolvan 75mg vs Lasolvan 30mg; Test type: Non-Inferiority or Equivalence — The assessment of relative bioavailability without molar mass adjustment (dose adjustment) was based upon two-sided 90% confidence intervals (CIs) for the ratios of the geometric means (test divided by reference) for the rate of absorption at steady state (Cmax ss/AUCss 0-24) using an acceptance range of 75%-133%; Adjusted Geometric Mean Ratio (%) = 76.55, 90% CI 2-sided [71.10 to 82.40], Standard Deviation 14.55 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV(%))
Statistical Analysis 2: Comparison: Lasolvan 60mg vs Lasolvan 30mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Adjusted Geometric Mean Ratio (%) = 100.46, 90% CI 2-sided [94.69 to 106.58], Standard Deviation 11.65 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV(%))
Statistical Analysis 3: Comparison: Lasolvan 75mg vs Lasolvan 60mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Adjusted Geometric Mean Ratio (%) = 75.69, 90% CI 2-sided [69.92 to 81.93], Standard Deviation 15.64 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV(%))

5. Secondary Outcome: Steady State Concentration of the Analyte in Plasma at the End of Dosing Interval
Description: Steady state concentration of the analyte in plasma at the end of dosing interval (Cmin ss)
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lasolvan 75mg | Lasolvan 60mg | Lasolvan 30mg
Number analyzed (Participants) | 23 | 23 | 23
ng/mL | 24.891 (39.355) | 22.740 (37.260) | 21.523 (40.803)

6. Secondary Outcome: Average Concentration of the Analyte in Plasma in the Time Interval of 0 to 24 h at Steady State
Description: Average concentration of the analyte in plasma in the time interval of 0 to 24 h at steady state (Cav ss)
Time Frame: as for outcome 1
Population: PK-BA set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lasolvan 75mg | Lasolvan 60mg | Lasolvan 30mg
Number analyzed (Participants) | 23 | 23 | 23
ng/mL | 49.254 (28.859) | 46.254 (28.292) | 44.621 (32.259)

7. Secondary Outcome: Time From Dosing to the Maximum Concentration of the Analyte in Plasma at Steady State
Description: Time from dosing to the maximum concentration of the analyte in plasma at steady state (tmax ss). For Lasolvan 30mg and Lasolvan 60mg, tmax ss was determined as tmax ss 0-12 and tmax ss 12-24.
Time Frame: as for outcome 1
Population: PK-BA set
Measure: Median (Full Range); unit: hours
Arm/Group | Lasolvan 75mg | Lasolvan 60mg | Lasolvan 30mg
Number analyzed (Participants) | 23 | 23 | 23
hours
  Tmax,ss,0-12h (N=0, 23, 23) | NA [NA to NA] — This was not determined for Lasolvan 75mg as dosing was once daily. | 1.00 [0.75 to 3.00] | 2.00 [0.75 to 3.00]
  Tmax,ss,12-24h (N=0, 23, 23) | NA [NA to NA] — This was not determined for Lasolvan 75mg as dosing was once daily. | 13.50 [12.75 to 16.00] | 14.00 [13.00 to 16.00]
  Tmax,ss,h (N=23, 0, 0) | 6.00 [2.00 to 12.00] | NA [NA to NA] — Tmax,ss was determined as tmax,ss 0-12 and tmax,ss 12-24 for Lasolvan 60mg as dosing was twice daily. | NA [NA to NA] — Tmax,ss was determined as tmax,ss 0-12 and tmax,ss 12-24 for Lasolvan 30mg as dosing was twice daily

8. Secondary Outcome: Peak-trough Fluctuation Between Minimum and Maximum Concentration of the Analyte in Plasma
Description: Peak-trough fluctuation between minimum and maximum concentration of the analyte in plasma (PTF)
Time Frame: as for outcome 1
Population: PK-BA set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lasolvan 75mg | Lasolvan 60mg | Lasolvan 30mg
Number analyzed (Participants) | 23 | 23 | 23
ng/mL | 0.994 (0.278) | 1.482 (0.322) | 1.483 (0.318)

9. Secondary Outcome: Peak-trough Swing
Description: Peak-trough swing (PTS) calculated as ((Cmax,ss - Cmin,ss / Cav,ss)*100)
Time Frame: as for outcome 1
Population: PK-BA set
Measure: Mean (Standard Deviation); unit: percentage of ng/mL
Arm/Group | Lasolvan 75mg | Lasolvan 60mg | Lasolvan 30mg
Number analyzed (Participants) | 23 | 23 | 23
percentage of ng/mL | 205.054 (82.703) | 313.106 (113.101) | 322.120 (135.222)

10. Secondary Outcome: Time Period When Concentration of the Analyte Exceeds Cav ss
Description: Time period when the concentration of the analyte exceeds Cav ss (T (C>Cav ss))
Time Frame: as for outcome 1
Population: PK-BA set
Measure: Median (Full Range); unit: hours
Arm/Group | Lasolvan 75mg | Lasolvan 60mg | Lasolvan 30mg
Number analyzed (Participants) | 23 | 23 | 23
hours | 10.500 [8.00 to 12.50] | 8.500 [5.75 to 10.00] | 7.750 [5.25 to 10.75]

11. Secondary Outcome: Plateau Time During Which Concentration of the Analyte in Plasma Exceeds 75% of Cmax ss
Description: Plateau time during which concentration of the analyte in plasma exceeds 75% of Cmax ss (T(C>75% Cmax ss))
Time Frame: as for outcome 1
Population: PK-BA set
Measure: Median (Full Range); unit: hours
Arm/Group | Lasolvan 75mg | Lasolvan 60mg | Lasolvan 30mg
Number analyzed (Participants) | 23 | 23 | 23
hours | 9.00 [0.00 to 13.00] | 2.25 [0.50 to 5.75] | 2.00 [0.50 to 5.25]

ADVERSE EVENTS:
Time Frame: From drug administration until the end of the consequent residual effect period (24 hours) for the treatment taken immediately before, 6 days
Arm/Group | Lasolvan 75mg | Lasolvan 60mg | Lasolvan 30mg
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.